CLINICAL TRIAL: NCT07232303
Title: The Effect of Cervical Stabilization Exercises on Pain, Mobility and Functionality in Temporomandibular Joint Dysfunction
Brief Title: The Effect of Cervical Stabilization Exercises in Temporomandibular Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Kumru Ateş, Assistant Professor, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KumruA
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Temporomandibular Joint Disorder
Keywords: Temporomandibular joint
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Stabilization Group (Experimental): cervical stabilization exercises, home exercises and patient education
  Interventions: Other: Cervical stabilization; Other: Home exercises; Other: Patient educating
- Control Group (Active Comparator): Home exercises and patient education
  Interventions: Other: Home exercises; Other: Patient educating

INTERVENTIONS:
Other: Cervical stabilization — Cervical range of motion exercises with craniocervical flexion, unilateral, bilateral and reciprocal shoulder flexion and abduction exercises, cervical isometric exercises with an exercise ball, unilateral, bilateral and reciprocal shoulder abduction when the exercise ball is between the wall and the head, and flexion exercises, exercise band and shoulder joint range of motion exercises with the exercise ball between the wall and the head were given to the study group. In the 3rd week, exercises were started with an exercise ball and elastic bands. All exercises were applied 3 times a day for 10 repetitions for 6 weeks.
  Arms: Cervical Stabilization Group
Other: Home exercises — The exercise program included mouth opening and closing against resistance, right-left lateral flexion movements, active mouth opening and closing, bilateral lateral flexion, protrusion, and retrusion. Stretching required the patient to perform the restricted movement, pushing their jaw toward the restricted direction with their hand, holding for 10 seconds, relaxing, and repeating. It also included self-massage in the form of stroking. All exercises were performed three times a day for 6 weeks, with 10 repetitions.
Other: Patient educating — The training content includes information about the disease, recommendations for a soft diet, avoidance of parafunctional habits, demonstration of diaphragmatic breathing, and notifications to ensure correct posture.

SUMMARY:
The purpose of this study is; to determine the efficacy of cervical stabilization exercises in the treatment of patients with temporomandibular joint disfunction

DETAILED DESCRIPTION:
Thirty patients diagnosed with temporomandibular joint dysfunction who were included in the study were randomly assigned to the 15-person control group and the study group. Patient training and home exercises for jaw joint were given to the control group while cervical stabilization exercise program was given to the study group. The program was administered by the patients for 6 weeks. Pre-treatment and post-treatment evaluations; active and passive maximum mouth openness, joint sounds, cervical range of motion, Visual Analogue Scale (VAS), Short Form Quality of Life Scale (Short Form-36), Tampa Kinesophobia Scale in Temporomandibular Disorders (TKS-TMD) and Pain Catastrophizing Scale (PCS), and the data obtained were analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Having a complaint of temporomandibular joint for more than 3 months.
* To be literate in Turkish.
* Having signed the Informed Consent Form.

Exclusion Criteria:

* -Those with active infection
* Presence of neurological, rheumatological and musculoskeletal problems that prevent exercise
* Vertebrobasilar artery insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
A Visual Analogue Scale | Change from initial assessment to 6 weeks after initial assessment
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.The TMJ pain caused by resting and activity of the individuals was measured using the Visual Analogue Scale (VAS) (0-10 interval scale) and was valued according to VAS.

SECONDARY OUTCOMES:
ROM TMJ | Change from initial assessment to 6 weeks after initial assessment.
  A 15 centimeter plastic ruler was used for ROM evaluation for TMJ. Depression of the active and passive mandible, lateral deviation (right and left), and protrusion were measured
Cervical ROM | Change from initial assessment to 6 weeks after initial assessment
  Cervical region ROM was evaluated with goniometer. Flexion, extension, rotation and lateral flexion (right and left) were measured. Each measurement was made 3 times and the mean value was recorded
Tampa Kinesiophobia Scale in Temporomandibular Disorders | Change from initial assessment to 6 weeks after initial assessment
  A 12-question questionnaire developed by Visscher and his friends, used in temporomandibular joint dysfunctions. 4-point Likert-type scoring is used. A total score of 12-48 is obtained. The higher the score a person receives, the higher the kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Yeniyüzyıl University Gaziosmanpaşa Hospital Dental Polyclinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No